CLINICAL TRIAL: NCT05566054
Title: A Multicenter, Randomized, Controlled Clinical Trial of Venetoclax, Azacytidine Combined With Chidamide for the Treatment of Newly Diagnosed Acute Monocytic Leukemia Patients That Are Ineligible for Intensive Chemotherapy
Brief Title: Venetoclax and Azacitidine Combined With Chidamide (VAC) for the Treatment of Newly Diagnosed Acute Monocytic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Jining Medical University (Other); The Second People's Hospital of Huai'an (Other); The First Affiliated Hospital of Bengbu Medical University (Other); Northern Jiangsu People's Hospital (Other); Affiliated Hospital of Nantong University (Other); Suzhou Hospital of Traditional Chinese Medicine (Other); Taizhou University (Other)
Responsible Party: Principal Investigator, Sheng-Li Xue, MD, Principal Investigator, The First Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZAMLM5
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Acute Monocytic Leukemia; Newly Diagnosed
Keywords: Chidamide; Azacitidine; Venetoclax
MeSH Terms: conditions — Leukemia, Monocytic, Acute | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Azacitidine; venetoclax

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VAC group (Experimental): Chidamide 10mg orally daily for 7 days (d1-d7), AZA 75mg/m2 daily for 7 days (d1-d7) and VEN orally once daily (100 mg d1, 200 mg d2, 400 mg d3-28); If the bone marrow assessment is CR/CRi/MLFS/PR/NR on the 21th-28th day in the first cycle, the second cycle of treatment will be started; If the bone marrow assessment is PR/NR, the patient needs to withdraw from the trial, If the bone marrow assessment is CR/CRi/MLFS, the patient will start post-remission therapy. For post-remission therapy, if the patients ineligible for intensive chemotherapy, continue with the same regimen until progression or recurrence of the disease, and the patients need to withdraw from the trial. If the patients were fit for intensive chemotherapy, patients will receive consolidation chemotherapy with other regimens or transplantation, and the patients needs to withdraw from the trial if progression or recurrence of the disease.
  Interventions: Drug: Chidamide; Drug: Azacitidine; Drug: Venetoclax
- VA group (Active Comparator): AZA 75mg/m2 daily for 7 days (d1-d7) and VEN orally once daily (100 mg d1, 200 mg d2, 400 mg d3-28); If the bone marrow assessment is CR/CRi/MLFS/PR/NR on the 21th-28th day in the first cycle, the second cycle of treatment will be started; If the bone marrow assessment is still PR/NR, the patient needs to enter VEN+AZA+Chidamide group. If the bone marrow assessment is CR/CRi/MLFS, the patient will start post-remission therapy. For post-remission therapy, if the patients ineligible for intensive chemotherapy, continue with the same regimen until progression or recurrence of the disease, and the patient needs to withdraw from the trial. If the patients fit for intensive chemotherapy, patients will receive consolidation chemotherapy with other regimens or transplantation, and the patient needs to withdraw from the trial if progression or recurrence of the disease.
  Interventions: Drug: Azacitidine; Drug: Venetoclax

INTERVENTIONS:
Drug: Chidamide — Chidamide 10mg orally daily for 7 days (d1-d7)
  Arms: VAC group
Drug: Azacitidine — azacytidine 75mg/m2 daily for 7 days (d1-d7)
Drug: Venetoclax — Venetoclax orally once daily (100 mg d1, 200 mg d2, 400 mg d3-28)

SUMMARY:
This study is to investigate the therapeutic efficacy and side effect of venetoclax, azacytidine combined with chidamide for newly diagnosed acute monocytic leukemia patients that are ineligible for intensive chemotherapy

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is one of the most aggressive blood cancers, with a very low survival rate and few options for patients who are unable to undergo intensive chemotherapy. Venetoclax in combination with hypomethylation agents or cytarabine has been approved by the Food and Drug Administration (FDA) for the treatment of patients with newly diagnosed AML unfit for intensive chemotherapy. However, resistance to venetoclax can be acquired through the upregulation of anti-apoptotic proteins in the BCL2 family, such as myeloid cell leukaemia 1 (MCL1). MCL1 plays a critical role in cell apoptosis regulation and high expression of MCL1 is observed in acute monocytic leukemia (AML-M5) . Chidamide, a newly designed selective histone deacetylase inhibitor, resulted in a decrease in the protein level of MCL1. This study is to investigate the therapeutic efficacy and side effect of venetoclax, azacytidine combined with chidamide for newly diagnosed AML-M5 patients that are ineligible for intensive chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Confirmation of acute monocytic leukemia( AML-M5) diagnosis by the French-American-British (FAB) Classification and/or characterized for expression of monocytic and myeloid differentiation markers, have a projected life expectancy of at least 12 weeks, previously untreated, and ineligible for treatment with intensive chemotherapy.

Patients must be considered ineligible for induction therapy defined by the following:

1. >= 60 years of age
2. >=18 to 59years of age with at least one of the following comorbidities:

   Any other comorbidity that the physician judges to be incompatible with intensive chemotherapy:

   (A)Eastern Cooperative Oncology Group (ECOG) performance status of 2 or 3. (B)Cardiac history of congestive heart failure requiring treatment or ejection fraction <= 50% or chronic stable angina.

   (C)Diffusing capacity of the lung for carbon monoxide (DLCO) <= 65% or forced expiratory volume during the first second (FEV1) <= 65%.

   (D)Creatinine clearance >= 30 mL/min to < 45 mL/min. (E)Moderate hepatic impairment with total bilirubin > 1.5 to <= 3.0 × upper limit of normal (ULN).
3. Must meet the laboratory requirements per the protocol.
4. Female participant must not be pregnant or breastfeeding and is not considering becoming pregnant or donating eggs during the study or for approximately 90 days after the last dose of study drug.
5. Female participants of childbearing potential must agree to use at least 1 protocol-specified method of birth control and male participants, if sexually active with female partner(s) of childbearing potential, must agree to practice the protocol-specified contraception.
6. Did not receive radiotherapy, chemotherapy, targeted therapy or hematopoietic stem cell transplantation within 4 weeks before enrollment;
7. Other comorbidities that are not suitable for intensive chemotherapy;
8. The patient refused to receive intensive chemotherapy;
9. Ability to understand and willing to sign the informed consent for this trial.

Exclusion Criteria:

1. Patients who are allergic to the study drug or drugs with similar chemical structures
2. Pregnant or lactating women, and women of childbearing age who do not want to practice effective methods of contraception
3. Active infection
4. Active bleeding
5. Patients with new thrombosis, embolism, cerebral hemorrhage, or other diseases or a medical history within one year before enrollment
6. Patients with mental disorders or other conditions whereby informed consent cannot be obtained and where the requirements of the study treatment and procedures cannot be met
7. Liver function abnormalities (total bilirubin > 1.5 times the upper limit of the normal range, ALT/AST > 2.5 times the upper limit of the normal range or patients with liver involvement whose ALT/AST > 1.5 times the upper limit of the normal range), or renal anomalies (serum creatinine > 1.5 times the upper limit of the normal value)
8. Patients with a history of clinically significant QTc interval prolongation (male > 450 ms; female > 470 ms), ventricular heart tachycardia and atrial fibrillation, II-degree heart block, myocardial infarction attack within one year before enrollment, and congestive heart failure, and patients with coronary heart disease who have clinical symptoms and requiring drug treatment
9. Urgery on the main organs within the past six weeks
10. Drug abuse or long-term alcohol abuse that would affect the evaluation results
11. Patients who have received organ transplants (excepting bone marrow transplantation)
12. Patients not suitable for the study according to the investigator's assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Composite Complete Remission Rate | At the end of Cycle 1 or 2 (each cycle is 28 days)
  The composite complete remission rate(complete remission plus complete remission with incomplete blood cell count recovery)
Overall response rate (ORR) | At the end of Cycle 1 or 2 (each cycle is 28 days)
  The overall response (completed remission without minimal residual disease, completed remission with incomplete blood count recovery, morphologic leukemia-free state and partial remission)

SECONDARY OUTCOMES:
Duration of Response (DOR) | 1 year
  It is measured the time from initial response to subsequent disease progression or relapse
Overall Survival (OS) | 1 year
  It is measured from the time of entry into this trial to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive
Progression-Free Survival (PFS) | 1 year
  It is measured from the time from randomization to progression or death
Adverse reactions in hematology | At the end of Cycle 1 (each cycle is 28 days)
  Record of adverse events in hematological system during and after VEN+AZA+Chidamide regimen induction (agranulocytosis days, PLT/RBC transfusion units)
Nonhematological adverse reactions | At the end of Cycle 1 (each cycle is 28 days)
  Record of adverse events in other organs or systmes during and after VEN+AZA+Chidamide regimen induction (infection and organ injury)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No